CLINICAL TRIAL: NCT05282628
Title: I-InTERACT Preterm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 315361
Record Dates: First submitted 2021-08-31; First posted 2022-03-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Pre-Term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Building Better Brains and Behavior program (B4 Preterm) (Experimental): Online learning modules completed sequentially and in conjunction with live coaching sessions led by a trained therapist.
  Interventions: Behavioral: Building Better Brains and Behavior program (B4 Preterm)

INTERVENTIONS:
Behavioral: Building Better Brains and Behavior program (B4 Preterm) — The program couples online learning modules with video conferencing sessions with a trained therapist to review skills and practice implementing the skills with live coaching. Online modules include didactic content, video clips of parents modeling the skills, and exercises. Parents will complete intervention modules sequentially in conjunction with scheduled 1:1 videoconference sessions with a trained therapist. Videoconference sessions with the therapist will be scheduled weekly, once parents have completed their modules. During these sessions, the therapist will review the online materials and provide active coaching to the parent on how to use the skills with their child (e.g., labeled praise, reflective responses). Each session follows a manualized therapy protocol to optimize content fidelity. Parents will be instructed to practice the parenting skills for 5 minutes each day to promote mastery in the home environment.

SUMMARY:
Open pilot of a brief online parenting-skills intervention for young children ages 3-8 who were born very preterm (< 32 weeks gestational age). Parent-child interactions, child behavior, parent functioning, and child white matter connectivity will be assessed pre- and post-intervention 10 weeks later.

DETAILED DESCRIPTION:
The investigators will modify I-InTERACT North to reflect United States language and culture and emphasize our focus on neural plasticity and development. The modified intervention will be renamed Building Better Brains and Behavior (B4 Preterm). Then, investigators will conduct a single-arm clinical trial to establish B4 Preterm's feasibility, acceptability and preliminary efficacy in improving child and family outcomes. Additionally, neuroimaging (MRI/DTI) will be collected pre- and post-intervention. The primary neuroimaging sequence will allow the investigators to examine associations between white matter injury and treatment response as well as changes in neural activation and connectivity pre- to post-treatment. An exploratory neuroimaging sequence will also be collected pre- and post-intervention. This exploratory sequence will serve as a backup for the primary sequence in case it is affected by significant motion and allow the investigators to test this sequence in young children.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: ages 3-8, inclusive
* Born at < 32 weeks gestational age
* Total T score of > 55 on the Child Behavior Checklist Total or Externalizing Behavior Scales OR Total T score of > 55 on the Eyberg Child Behavior Inventory total problem- or total intensity-scale OR documented behavioral problems noted in medical chart and parent endorses current concerns about child's behaviors
* Language: English must be the primary spoken language in the home

Exclusion Criteria:

Caregiver must be 18 years or older to participate in the intervention. Participant will be excluded from the study if the child does not reside with the caregiver at least half-time; the caregiving situation is not stable (i.e., there must be no scheduled custody hearings); English is not the primary language spoken in the home. Additionally, caregivers with a psychiatric hospitalization in the past year will be ineligible to participate. Children with certain types of metal in their heads will be unable to participate in the MRI portion but will be able to participate in the intervention and complete pre- and post-intervention questionnaires.

Ages: 36 Months to 96 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | Week 1
  Child Behavior
Eyberg Child Behavior Inventory (ECBI) | Week 10
  Child Behavior
Child Behavior Checklist | Week 1
  Child Behavior
Child Behavior Checklist | Week 10
  Child Behavior
Behavior Rating Inventory of Executive Functions-2 | Week 1
  Executive Function Behaviors
Behavior Rating Inventory of Executive Functions-2 | Week 10
  Executive Function Behaviors
Center for Epidemiologic Studies Depression Scale (CES-D) | Week 1
  Caregiver Depression; Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Center for Epidemiologic Studies Depression Scale (CES-D) | Week 10
  Caregiver Depression; Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Adverse Childhood Experiences Scales (ACES) | Week 1
  Caregiver Stress; Scores range from 0 to 10, with higher scores indicating a higher risks for developing later health problems.
Adverse Childhood Experiences Scales (ACES) | Week 10
  Caregiver Stress; Scores range from 0 to 10, with higher scores indicating a higher risks for developing later health problems.
Pediatric Quality of Life Inventory (PedsQL) | Week 1
  Child functioning and quality of life
Pediatric Quality of Life Inventory (PedsQL) | Week 10
  Child functioning and quality of life
Dyadic Parent Child Interaction Coding System (DPICS) | Week 1
  Parenting Behaviors
Dyadic Parent Child Interaction Coding System (DPICS) | Week 10
  Parenting Behaviors
Satisfaction Survey | Week 10
  Satisfaction with Intervention

SECONDARY OUTCOMES:
Multi-shell diffusion sequence | Week 1
  Neuroimaging-MRI/DTI
Multi-shell diffusion sequence | Week 10
  Neuroimaging-MRI/DTI
3D-T1 weighted sequences | Week 1
  Neuroimaging-MRI/DTI
3D-T1 weighted sequences | Week 10
  Neuroimaging-MRI/DTI
3D T2- weighted sequence | Week 1
  Neuroimaging-MRI/DTI
3D T2- weighted sequence | Week 10
  Neuroimaging-MRI/DTI
Resting state fMRI sequence | Week 1
  Neuroimaging-MRI/DTI
Resting state fMRI sequence | Week 10
  Neuroimaging-MRI/DTI

CONTACTS AND LOCATIONS:
Overall Officials: Shari L Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States